CLINICAL TRIAL: NCT05471791
Title: Development of a Concussion Management Platform for Children and Youth: Bridging the Gap Between Research and Practice
Brief Title: Development of a Concussion Management Platform for Children and Youth
Acronym: Back2PlayApp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Natural Sciences and Engineering Research Council, Canada (Other); McMaster Children's Hospital (Other); Montreal Children's Hospital of the MUHC (Other); Hamilton-Wentworth Catholic District School Board (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRP 538798-19
Record Dates: First submitted 2022-04-14; First posted 2022-07-25 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-06

CONDITIONS: Concussion, Brain
Keywords: youth or children; mHealth
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Randomized control trial comparing treatment (use of mobile App) to usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App group (Experimental): Participants will use the Back2Play App to support them in following the guidelines for recovery from concussion
  Interventions: Device: Back2Play App
- Usual Care (No Intervention): Participants will receive usual care which often means they are provided concussion recovery guidelines in handout format and receive whatever follow up is deemed necessary by treating physician

INTERVENTIONS:
Device: Back2Play App — This App uses the Apple watch to monitor activity level and heart rate and combines this with self reported symptoms and stage of recovery to send notifications, suggestions and provide resources to help participants adhere to the guidelines.
  Arms: App group

SUMMARY:
This multi-centred, randomized controlled trial will evaluate the effectiveness of a pilot tested mobile device Application built to guide youth in recovery from concussion. The Back2Play App was developed based on the published and researched CanChild Return to Activity (RTA) and Return to School (RTS) guidelines, which outline graduated steps in returning to play and school for youth after a concussion. It is hypothesized that participants who use the App will have better outcomes from concussion, primarily less reinjury during the vulnerable period throughout their recover up to 3 months after concussion. They may also experience reduced frequency and severity of symptoms and recover more quickly from their concussion.

DETAILED DESCRIPTION:
Children 10- 18 years of age will be recruited from Emergency departments in Hamilton, Ontario and Montreal, Quebec as well as from community physicians, school boards and sporting organizations. All participants will be randomized to either the App (intervention) group or to Usual care (control) group.

Those in the App group will be loaned an Apple watch (and iPhone if they don't have one). The App is designed to monitor self-reported symptoms and stages of recovery and combine these results with their activity and heart rate data collected by the watch. Notifications are sent through the App based on this data that may help youth adhere to the Return to Activity and Return to School (RTA/RTS) guidelines. Participants will fill out symptom surveys in the App up to 3 times daily, record their physical and cognitive activities and assign themselves a stage of recovery; RTA 1-6, RTS 1-5. The homepage of the App reminds them of what stage they are in of RTA and RTS as well as how much light, moderate and vigorous activity is encouraged for their individual stage of recovery. They will receive notifications about activity level and heart rate if these go outside the recommended limits. App users will also receive motivational statements and encouragement.

The control group will receive usual care with the approach provided in health care systems in their community. This often involves a handout with some type of graduated rest and return to play advice. These participants will complete the initial Post Concussion Symptom Scale at their entry into the study and will be sent daily symptom and activity surveys by our secure data capture system (REDCap) to complete. They will also be asked to self-select their stage of concussion recovery daily for both activity and school.

All participants will be scheduled for a zoom interview after their symptoms are gone, or 3 months after enrolling for those who do not achieve full recovery during the study. They will be asked questions about: 1) their understanding and experience with concussion recovery, 2) whether they experienced another head injury and 3) if those who used the App liked it and found it helpful. 3 months after study completion, participants will receive another survey asking if they have experienced any additional head injuries. Those using the App will be given the System Usability Scale (SUS) to objectively rate the App for potential future commercialization.

All data will be analyzed as discussed in the study protocol. Data may also be used fill in the architecture of a machine learning algorithm running in the background of the Back2Play App to use in predicting RTA/RTS stages for participants in future iterations of the App.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed concussion
* symptomatic
* within 4 weeks of diagnosis

Exclusion Criteria:

* developmental delay
* significant brain injury requiring resuscitation, admission to PCCU or surgical intervention
* multisystem injury

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 181 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Rate of re-injury | Surveyed 3 months after completion of study (6 months maximum from enrollment)
  Survey-report on whether another concussion has occurred. Yes/No response
Change in number and severity of Post-concussive symptoms (PCSS) | Throughout the study until recovered or up to a maximum of 3 months after enrolment
  Daily surveys of 22 concussion symptoms (1symptom/0 no symptoms) for # of symptoms. Included in these surveys is report of symptom changes (gone, better, same or worst) that will help to evaluate changes by stage of recovery and over the course of recovery.

SECONDARY OUTCOMES:
Time to recovery from concussion | Through study completion, an average of 1 month, up to 6 months post-enrollment
  Measurement of time from injury to when youth have recovered (return to activity stage 6/return to school stage 5)
System Usability Scale (SUS) (for the App group only) | upon completion of study (max 3 months post enrollment)
  10 item questionnaire using a Likert scale with five response options for measuring usability of a system (App) 1=strongly disagree 5= strongly agree; Scores are converted to an overall percentage with 70% and above a good score

CONTACTS AND LOCATIONS:
Overall Officials: Carol A DeMatteo, MSc, Principal Investigator — McMaster University FHS
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Montreal Children's Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 9 months and ending 36 months after article publication.
Access Criteria: Proposals for data analysis will be considered if there is a methodologically sound request. All requests should go through the PI dematteo@mcmaster.ca

REFERENCES:
- [Background] DeMatteo CA, Lin CA, Foster G, Giglia L, Thabane L, Claridge E, Noseworthy MD, Hall GB, Connolly JF. Evaluating Adherence to Return to School and Activity Protocols in Children After Concussion. Clin J Sport Med. 2021 Nov 1;31(6):e406-e413. doi: 10.1097/JSM.0000000000000800. PMID 31876794
- [Background] DeMatteo C, Bednar ED, Randall S, Falla K. Effectiveness of return to activity and return to school protocols for children postconcussion: a systematic review. BMJ Open Sport Exerc Med. 2020 Feb 24;6(1):e000667. doi: 10.1136/bmjsem-2019-000667. eCollection 2020. PMID 32153982
- [Background] DeMatteo C, Randall S, Falla K, Lin CY, Giglia L, Mazurek MF, Koelink E. Concussion Management for Children Has Changed: New Pediatric Protocols Using the Latest Evidence. Clin Pediatr (Phila). 2020 Jan;59(1):5-20. doi: 10.1177/0009922819879457. Epub 2019 Oct 18. PMID 31625406
- [Background] DeMatteo CA, Randall S, Lin CA, Claridge EA. What Comes First: Return to School or Return to Activity for Youth After Concussion? Maybe We Don't Have to Choose. Front Neurol. 2019 Jul 23;10:792. doi: 10.3389/fneur.2019.00792. eCollection 2019. PMID 31396150
- See also: CanChild Research centre website with Back2Play App study updates — https://www.canchild.ca/en/research-in-practice/current-studies/the-back2play-app-study
- See also: CanChild published Return to Activity and Return to School guidelines for Youth recovering from concussion — https://canchild.ca/en/resources/249-concussion-mild-traumatic-brain-injury-guideline-brochures

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05471791/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05471791/ICF_001.pdf